CLINICAL TRIAL: NCT02918500
Title: Effect of Pre-operative Nicotine Replacement Therapy on Peri-operative Complications and Long-term Abstinence: A Pilot Placebo-controlled Trial in Patients Undergoing Coronary Artery Bypass Surgery (CABG)
Brief Title: Effect of Pre-op NRT on Peri-operative Complications and Long-term Abstinence: A Pilot Trial in Patients Undergoing CABG Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to recruitment challenges.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160696-01H
Record Dates: First submitted 2016-09-06; First posted 2016-09-29 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Smoking Cessation
Keywords: Coronary Artery Bypass Surgery (CABG); Nicotine Replacement Therapy (NRT)
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Participants will receive 3 weeks of inactive NRT patches.
- Active (Active Comparator): Participants will receive 3 weeks of active NRT patches
  Interventions: Drug: Nicoderm Patch

INTERVENTIONS:
Drug: Nicoderm Patch — Nicotine replacement therapy patch
  Arms: Active

SUMMARY:
This study will determine whether or not patients who use a Nicotine Replacement Therapy (NRT) patch prior to their by-pass surgery are more likely to be smoke-free 6 months after their surgery and have fewer post-operative complications

DETAILED DESCRIPTION:
The aim of this project is to

1. To determine if pre-operative, (short-term) NRT, 1 to 3 weeks before surgery, improves the long-term quit rates among smokers undergoing elective CABG surgery.
2. To determine the effect of pre-operative NRT on perceived stress and symptoms of nicotine withdrawal at the time of surgery.
3. To assess, retroactively, the impact of pre-operative cessation on peri-operative complications such as infection rates, respiratory failure, myocardial infarction, stroke, sepsis, shock and prolonged hospital stay.

We therefore hypothesize that if NRT is given to smokers during the pre-admission period (1-3 weeks prior to surgery), they are more likely to be biochemically abstinent from cigarette smoking 6 months after hospitalization and will experience fewer peri-operative complications

To assess these measures, we have designed a single site, double-blinded randomized controlled trial at the University of Ottawa Heart Institute (UOHI). Patients who are identified as a smoker at their initial visit to the PAU will undergo a baseline assessment and be randomly assigned (1:1) to either active or placebo 21mg NRT patch. They will wear the patch from that baseline visit until the day of their surgery at UOHI. Following their surgery, they will receive a follow up phone call at 1 and 6 months post-discharge. They will complete a series of short questionnaires to assess their smoking status, stress levels and nicotine withdrawal symptoms. Those who identify themselves as being smoke-free will be asked to complete a carbon monoxide breathing test to chemically validate their smoking status. The study protocol will be reviewed by the Research Ethics board at UOHI and all participants will provide written informed consent prior to undertaking any study activities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently smoking >5 cigarettes/day for the past 30 days; there is no evidence that NRT is useful in those who smoke <5cpd.
2. Patient is able to participate and willing to provide informed consent; participants will need to follow directions and adhere to the medication usage instructions as outlined in the informed consent document.
3. Patients is willing to be contacted by phone for follow up at 1 month and 6 months post-discharge; these time points will assess our final outcome of cessation at 6 months post-discharge.

Exclusion Criteria:

1. Patient is scheduled for surgery in < 7 days; most patients need to be using NRT consistently for 2 weeks for it to be fully effective.
2. Patient is currently using a smoking cessation product (i.e. nicotine containing patch, gum, inhaler, lozenge, spray or nicotine containing electronic cigarette, varenicline, buproprion) or has used a smoking cessation aid consistently for more than 72 consecutive hours with the intent to reduce cigarette consumption or quit smoking within 30 days of the baseline Pre-admission Unit (PAU) visit; this will ensure the effects of the study patches will be assessed without any contamination from other cessation products.
3. Patient is willing to refrain from using any other cessation products (nicotine containing patch, gum, inhaler, lozenge, spray, nicotine containing electronic cigarette, varenicline, buproprion) prior to surgery; this will allow us to track the usage and side effects with the study patches.
4. Patient is allergic to the adhesive on the nicotine replacement therapy patch.
5. Patient is unable to read and understand English or French; study materials will only be supplied in these two languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pipe, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Active
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 65 [54 to 76] | 70 [57 to 83] | 68.5 [54 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Carbon Monoxide (CO) Confirmed Abstinence at the Time of Surgery
Description: To determine if pre-operative, (short-term) NRT, 1 to 3 weeks before surgery, improves the long-term quit rates among smokers undergoing elective CABG surgery
Time Frame: At the time of CABG surgery (will vary with all participants based on their surgical date) and at each follow up visit (1 month and 6 month post-op)
Population: Study terminated due to recruitment challenges. Only 4 participants were recruited and therefore there was not enough data to warrant analysis.
Arm/Group | Placebo | Active
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Effect of Pre-operative NRT on Perceived Stress and Symptoms of Nicotine Withdrawal at the Time of Surgery
Description: Measured by the perceived stress scale (PSS-14)
Time Frame: At the time of surgery and each follow up visit (1 & 6 months post-op)
Population: Due to a small sample size recruited for this trial, the follow up data was not assessed within either group
Arm/Group | Placebo | Active
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: The Impact of Pre-operative Cessation on Peri-operative Complications Such as Infection Rates, Respiratory Failure, Myocardial Infarction, Stroke, Sepsis, Shock and Prolonged Hospital Stay.
Description: Participants will be asked about any post-operative complications and a retrospective chart review will be completed for all participants.
Time Frame: assessed at the 1 and 6 month post-op follow up visits
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 8 months (recruitment start to recruitment termination). Participants were monitored for adverse events during their 3 week intervention period.
Description: Adverse events were reported by the participants to the Research Coordinator. Participants were directly asked about adverse events during each study contact.
Arm/Group | Placebo | Active
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Study was terminated early due to recruitment challenges; only 4 participants were recruited. The data for these 4 participants will not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT02918500/Prot_000.pdf